CLINICAL TRIAL: NCT06556069
Title: Peer Support Enhanced Behavioral Crisis Response Teams in the Emergency Department
Brief Title: Clinical Trial of Peer Support in the ED (PCORI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000038473; BPS-2022C3-30381 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Psychomotor Agitation; Behavioral Disorder
Keywords: Agitation; Peer Support
MeSH Terms: conditions — Psychomotor Agitation; Mental Disorders

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge, cluster randomized study design that evaluates the impact of the PACT intervention. Our unit of randomization is at the cluster (i.e., ED site) level. A sample of five ED sites will complete the stepped-wedge cluster randomized trial with six time periods (including the baseline), five steps, and each site randomized from control to intervention at each step. The trial will be conducted over three years, with each period duration being six months.
Masking Description: We will not utilize masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard of care will occur during the baseline/pre-implementation phase and no quality improvement programs or interventions related to agitation management will occur during this time period.
- PACT Implementation (Experimental): Implementation of the PACT intervention. After a site is randomized to implement PACT, trained peers will be assigned to work ED shifts alongside the structured code team. ED patients with behavioral needs will receive peer-led TIC, including empathic listening, therapeutic relationship building, understanding of patient needs and goals for the visit, and informing of patients and family about the evaluation process in real-time.
  Interventions: Other: Peer-Support Enhanced Agitation Code Team (PACT)

INTERVENTIONS:
Other: Peer-Support Enhanced Agitation Code Team (PACT) — PACT will address systems challenges experienced by staff, safety threats to ED patients with mental illness and substance use disorders, and known structural biases against marginalized individuals during decisions in use of restraints for behavioral crises in the ED.
  The PACT intervention includes a peer support service component to deliver patient-centered, trauma-informed, culturally sensitive care to patients presenting with behavioral complaints in the ED and experiencing distress.
  Arms: PACT Implementation

SUMMARY:
The purpose of this study is to conduct a clinical trial that tests the acceptability, fidelity, and feasibility of a peer support modified intervention for agitation management within the emergency department.

DETAILED DESCRIPTION:
The purpose of this study is to address the increasing burden of behavioral crises and agitation in the Emergency Department (ED). There are multiple significant gaps in patient centered care for agitation management and use of restraints in the context of behavioral crises, leading to increased patient risks and reduced workplace safety. Through expanding our previous Agitation Code Team (ACT) protocol with the addition of peer support workers, we plan to develop a peer-support enhanced agitation code team (PACT). The PACT will address systems challenges experienced by staff, safety threats to ED patients with mental illness and substance abuse disorders and reduce known structural biases in marginalized patient populations during restraint/sedation decision making. Additionally, peer support workers delivery of trauma informed care is the key mechanism for mitigating bias in agitation management.

This study will build on our team's extensive experience in using a patient-centered approach for investigating best practices in management of agitation in the ED. Thus, we propose a patient centered, trauma informed, structured team-based care delivery approach through the use of a multi-level, multi-component peer-support enhanced agitation code team (PACT) intervention. PACT will address systems challenges experienced by staff, safety threats to ED patients with mental illness and substance use disorders, and known structural biases against marginalized individuals during decisions in use of restraints for behavioral crises in the ED. We hypothesize that the PACT intervention will improve patient outcomes related to behavioral crisis (i.e., reduction in use of restraints, engagement to follow-up care, decrease in repeat ED visits) and improve patient experience of behavioral acute care in the ED for patients presenting with behavioral health chief complaints, especially those from racial/ethnic minority groups and historically marginalized populations compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English-speaking
* Arrives to one of the Yale-New Haven Health emergency departments (Yale-New Haven [York Street & St. Raphael's], Greenwich, Bridgeport, Lawrence & Memorial, and Westerly campuses)
* Presents with a behavioral-related chief complaint (inclusive of neurocognitive, substance use/intoxication, mental health and other behavioral related presentations) as well as additional individuals at risk of developing agitation defined via a score of >2 on the Brøset Violence Checklist

Exclusion Criteria:

* Pregnant women, minors (<18 years old), prisoners, and institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57870 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Restraint Use | Up to 1 day
  Our primary outcome will be rates of Restraint Use, which will be the percent of patients with a behavioral health chief complaint or at risk for agitation who receive either a physical restraint or chemical restraint (defined as intramuscular administration of a sedative) order during an ED visit, measured as a rate per 1,000 ED visits.

SECONDARY OUTCOMES:
Agitation Symptom Level | Up to 1 day
  Levels and symptoms of agitation during an ED visit will be measured by the Brøset Violence Checklist (BVC), a validated risk assessment tool used to predict violent behavior within a 24-hour period based on presence or absence of patient behaviors and characteristics.
  Minimum score = 0 and maximum score = 6. Interpretation as follows: 0 score indicates a small/low risk of violence, a score of 1-2 indicates moderate risk of violence, and a score greater than 2 indicates high risk of violence and a need to develop a plan to manage patient's violence.

CONTACTS AND LOCATIONS:
Overall Officials: Ambrose Wong, MD, MSEd, MHS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital Health System, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nath B, Desai R, Cook JM, Dziura JD, Davis-Plourde K, Youins R, Guy K, Pavlo AJ, Smith PE, Smith PD, Kangas K, Heckmann R, Hart L, Powsner S, Sevilla M, Evans M, Kumar A, Faustino IV, Hu Y, Bellamy C, Wong AH. Peer support enhanced behavioural crisis response teams in the emergency department: protocol for a stepped-wedge cluster-randomised controlled trial. BMJ Open. 2025 Jun 8;15(6):e103775. doi: 10.1136/bmjopen-2025-103775. PMID 40484432